CLINICAL TRIAL: NCT02616419
Title: External Cold and Vibration Stimulation (Buzzy® Device) VS Topical Anesthetic Cream for Procedural Pain Management in Children Undergoing Needle-Related Procedures in the Emergency Department : A Randomized Controlled Non-Inferiority Trial
Brief Title: External Cold and Vibration Stimulation (Buzzy®) for Procedural Pain Management in Children Undergoing Needle-Related Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Ariane Ballard, PhD Student, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-1405
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Child; Pain Due to Certain Specified Procedures
Keywords: Emergency Department; Procedural pain; Procedural anxiety; Needle-related procedures; Clinical Nursing Research; Nursing practice; Non-pharmacological method
MeSH Terms: conditions — Emergencies; Pain, Procedural | interventions — Maxilene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Buzzy® device (Experimental): Just before the needle-related procedure, the Buzzy®, combining an ice pack and vibration integrated to a plastic bee, will be applied 5 cm above the needle insertion site and will be maintained in place throughout the painful procedure.
  Interventions: Device: Buzzy® device
- Maxilene® (Lidocaine liposomal 4%) (Active Comparator): Maxilene® topical anaesthetic cream will be applied 30 minutes before the needle-related procedure at the insertion site.
  Interventions: Drug: Maxilene® (Lidocaine liposomal 4%)

INTERVENTIONS:
Device: Buzzy® device — Just before the needle-related procedure, the Buzzy®, combining an ice pack and vibration integrated to a plastic bee, will be applied 5 cm above the needle insertion site and will be maintained in place throughout the painful procedure.
  Arms: Buzzy® device
Drug: Maxilene® (Lidocaine liposomal 4%) — Maxilene® topical anaesthetic cream will be applied 30 minutes before the needle-related procedure at the insertion site.
  Arms: Maxilene® (Lidocaine liposomal 4%)

SUMMARY:
Since the late 1980s, several studies focused on pediatric procedural pain and show that it still underevaluated and undertreated, especially in the Emergency Department (ED). Needle-related procedures are the most important source of pain and anxiety and children. Since it is impossible to completely eliminate the pain and anxiety experienced by children during painful procedures, use of non-pharmacological and/or pharmacological interventions might be beneficial. Most methods used for relief of procedural pain and anxiety for children require time or extra staff, which represent barriers to their implantation in the ED. An easy-to-use and rapid non-pharmacological intervention could overcome these constraints and optimize procedural pain and anxiety relief in children undergoing a needle-related procedure.

The primary objective of this study is to determine if a device combining cold and vibration (Buzzy®) is non-inferior (no worse) than a topical anesthetic cream (lidocaine liposomal 4%) for procedural pain management in children undergoing needle-related procedures in the ED.

Investigators strongly believe that the use of the Buzzy® device in the ED will improve significantly the pain and anxiety felt by children undergoing needle-related procedures. Since EDs are usually chaotic and very busy, an easy-to-use and rapid non-pharmacological intervention like the Buzzy®, will surely be adopted by the nursing personnel as a useful tool for procedural pain. Given this knowledge, the investigators feel that this randomized controlled trial will have the potential to improve nursing practice and optimize painful experiences of children undergoing needle-related procedures.

DETAILED DESCRIPTION:
Since the 1980s, several researches focused on paediatric procedural pain to learn more about its nature, its causes, its consequences, its assessment and treatment. However, decades later, it is still undervalued and undertreated, especially in the Emergency Department (ED). Thus, children experience a high level of pain and anxiety in the ED during painful procedures, which could be due to multiple factors: lack of knowledge regarding pain management interventions, lack of time, work overload, limited space and interruption in the continuity of care.

Needle-related procedures (venipuncture, IV access, s/c, IM) are the most important sources of pain and distress in children. A study shows that only 31% of children benefit from procedural pain management during the insertion of an IV access and less than 1% during a venipuncture. Inadequate procedural pain and anxiety relief in children is not without consequences. These effects may be physiological, psychological and emotional and can have long-term impact. Since it is impossible to completely eliminate the pain and anxiety experienced by children during needle-related procedures, relief through non-pharmacological and/or pharmacological interventions is essential.

Most relief methods of procedural pain and anxiety available for children require much time or staff, which represent barriers regarding their implantation in the ED. The use of a rapid and easy-to-use non-pharmacological intervention could overcome these constraints and optimize procedural pain and anxiety relief in children. In 2009, a new device (Buzzy®), combining cold (ice wings) and vibration (bee's body), was developed in the USA for the relief of pediatric procedural pain. This device relies on the Gate Control Theory as well as diffuse noxious inhibitory control for the modulation of pain response (Baxter et al., 2009). Efficacy of the Buzzy® device in pediatric patients in the ED has only been evaluated in two studies up to this date. Both studies showed significant results regarding control of post-procedural pain and post-procedural anxiety. So far, no study has been conducted in Canada and none has compared the effects of Buzzy. Since the 1980s, several researches focused on pediatric procedural pain to learn more about its nature, its causes, its consequences, its assessment and treatment. However, decades later, it is still undervalued and undertreated, especially in the Emergency Department (ED). Thus, children experience a high level of pain and anxiety in the ED during painful procedures, which could be due to multiple factors: lack of knowledge regarding pain management interventions, lack of time, work overload, limited space and interruption in the continuity of care.

Needle-related procedures (venipuncture, IV access, s/c, IM) are the most important sources of pain and distress in children. A study shows that only 31% of children benefit from procedural pain management during the insertion of an IV access and less than 1% during a venipuncture. Inadequate procedural pain and anxiety relief in children is not without consequences. These effects may be physiological, psychological and emotional and can have long-term impact. Since it is impossible to completely eliminate the pain and anxiety experienced by children during needle-related procedures, relief through non-pharmacological and/or pharmacological interventions is essential.

Most relief methods of procedural pain and anxiety available for children require much time or staff, which represent barriers regarding their implantation in the ED. The use of a rapid and easy-to-use non-pharmacological intervention could overcome these constraints and optimize procedural pain and anxiety relief in children. In 2009, a device (Buzzy®), combining cold (ice wings) and vibration (bee's body), was developed in the USA for the relief of pediatric procedural pain. This device relies on the Gate Control Theory as well as diffuse noxious inhibitory control for the modulation of pain response (Baxter et al., 2009). The few study that have evaluated its efficacy presents several limitations, such as small sample size and absence of intervention in control group. To date, no study has been conducted in Canada and none has compared its effects with the gold standard intervention for needle-related procedures, the topical anesthetic cream.

Objective:

The primary aim of this study is to determine if a device combining cold and vibration (Buzzy®) is non-inferior (no worse) than lidocaine liposomal 4% for procedural pain management in children undergoing needle-related procedures in the ED.

Methods:

Design: This study is a two-arm, randomized, controlled, non-inferiority trial. Setting: Pediatric ED in a university health center in Montreal. Inclusion criteria: Investigators will include children: 1) Ages from 4-17 years old; 2) Visiting the ED; 3) Requiring a needle-related procedure (venipuncture or IV catheter insertion); 4) Understanding and speaking either French or English; 5) Having at least one parent (or legal guardian) who understands, read and talks in French or English. Exclusion criteria: Investigators will exclude children with: 1) A neuro-cognitive impairment that precludes informed consent and/or assent, 2) An inability to self-report pain, 3) A critical or unstable health. Interventions: Arm 1 (Buzzy® device): Just before the needle-related procedure, the Buzzy® device (combining an ice pack and vibration integrated to a plastic bee) will be applied 5 cm above needle insertion site and will be maintained in place throughout the painful procedure. Arm 2 (lidocaine liposomal 4%): The topical anesthetic cream will be applied 30 minutes before the needle-related procedure on the insertion site. Randomization and Allocation: A independent biostatistician will generate the sequence of randomization stratified by age (4-7; 8-12; 13-17) and using permuted block sizes for each stratum. Enrolled participants will be randomly assigned to one of the two arms with a 1:1 allocation ratio. Sample size: Using a non-inferiority margin of 0.7 on a scale 0 to 10 for mean per-procedural pain, a total of 380 participants (190/group) will be necessary to achieve a power of 90% at the one-sided 5% significance. Primary outcome: The primary outcome will be the mean per-procedural pain scores on the Color Analogue Scale (CAS). Secondary outcomes: a) Mean per-procedural pain scores on Faces-Pain Scale Revised (FPS-R), b) Mean level of per-procedural distress using the Procedure Behavior Check List (PBCL) and the Children's Fear Scale (CFS), c) Memory of pain 24 hours after the needle-related procedure on the FPS-R. d_ Proportion of children with success of the needle-related procedure at first attempt, e) Self-reported levels of satisfaction of children, parents and nurses with questionnaires previously developped by our team. Analyses: All analyses will be performed under both intention-to-treat and per-protocol principles. Regarding the primary outcome, the mean difference in pain scores between the experimental group ( Buzzy® device) and the control group (lidocaine liposomal 4%) along with its lower confidence limit will be calculated. If this limit lies within (-∞,0.7), then the null hypothesis of inferiority will be rejected in favor of the alternative hypothesis at the 5% significance level. A similar approach will be used for the secondary outcomes (a, b, c). Proportion of children with success of the procedure at first attempt will be compared using a chi-square test. Descriptive statistics will be used to report data on satisfaction. ANCOVA will be performed on covariate to increase statistical power. Subgroups analyses will be performed according to age groups (4-7; 8-12; 13-17).

Relevance :

This proposed work will be the first RCT in Canada to assess the efficacy of the Buzzy® device for procedural pain and anxiety relief in children undergoing needle-related procedure. Very few studies of pharmacological and non-pharmacological interventions exist, but no intervention have been identified to be optimal for pain and anxiety management in the context of an ED. Investigators strongly believe that the use of the Buzzy® device in children undergoing needle-related procedures would optimize nursing practice and improve pain and anxiety experienced by children during their visit to the ED.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 4 and 17 years old
* Visiting the Emergency Department
* Requiring a venipuncture or IV catheter insertion
* Able to understand and speak French or English
* Having at least one parent who can understand, read and talk in French or English

Exclusion Criteria:

* Neuro-cognitive disability that precludes patients from assenting and participating to the study
* Inability to self-report pain
* Critical or unstable health status

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Mean per-procedural pain scores | T-3: Immediately after the-needle-related procedure
  The per-procedural pain intensity will be assess immediately after the needle-related procedure using the Color Analogue Scale (CAS) (self-report scale).

SECONDARY OUTCOMES:
Mean per-procedural pain scores | T-3: Immediately after the needle-related procedure
  The per-procedural pain intensity will be assess immediately after the needle-related procedure using the Faces Pain Scale-Revised (FPS-R) (self-report scale).
Mean level of per-procedural distress | T-2: During the needle-related procedure
  The level of per-procedural distress will be assess during the needle-related procedure using the Procedure Behavior Check List (PBCL) (observational scale).
Mean level of per-procedural distress | T-3: Immediately after the needle-related procedure
  The level of per-procedural distress will be assess immediately after the needle-related procedure using the Children's Fear Scale (CFS) (self-report scale).
Satisfaction regarding the use of the Buzzy® device | T-4: 15 minutes after the needle-related procedure
  The satisfaction of the nurses, children and parents regarding the use of the Buzzy® device will be assess after the needle-related procedure with questionnaires previously developped by the investigators.
Memory of pain (mean post-procedural pain scores 24 hours after the procedure) | T-5: 24 hours after the needle-related procedure
  The memory of pain will be assess 24 hours after the needle-related procedure using the Faces-Pain Scale-Revised (FPS-R) (self-report scale).
Proportion of participants with success of the needle-related procedure at the first attempt | T-3: Immediately after the needle-related procedure
  The success of the needle-related procedure at first attempt will be assess using dichotomized (yes/no) clinical data immediately after the needle-related procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Ballard, PhD Student, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ballard A, Khadra C, Adler S, D Trottier E, Bailey B, Poonai N, Theroux J, Le May S. External cold and vibration for pain management of children undergoing needle-related procedures in the emergency department: a randomised controlled non-inferiority trial protocol. BMJ Open. 2019 Jan 15;9(1):e023214. doi: 10.1136/bmjopen-2018-023214. PMID 30782698